CLINICAL TRIAL: NCT03054519
Title: Improve PAD Performance With Metformin: The PERMET Trial
Brief Title: Improve PAD PERformance With METformin
Acronym: PERMET
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Northwestern University (Other)
Responsible Party: Principal Investigator, Mary McDermott, Professor of Medicine at Northwestern University Feinberg School of Medicine, Northwestern University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: STU00203784
Record Dates: First submitted 2017-02-13; First posted 2017-02-15 (Actual); Last update posted 2025-08-26 (Actual); Status verified 2025-08

CONDITIONS: Peripheral Artery Disease
MeSH Terms: conditions — Peripheral Arterial Disease | interventions — Metformin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Metformin (Active Comparator): Metformin daily
  Interventions: Drug: Metformin
- Placebo (Placebo Comparator): Placebo daily for six months.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Metformin — Participants will be prescribed up to 2,000 mgs daily of metformin
  Arms: Metformin
Drug: Placebo — Placebo pills will appear identical to the metformin to maintain blinding of participants and investigators.
  Arms: Placebo

SUMMARY:
The PERMET trial will determine whether metformin daily for six months improves six-minute walk performance in individuals with peripheral artery disease compared to placebo.

ELIGIBILITY:
Inclusion Criteria:

All participants will have PAD. PAD will be defined as follows:

* First, an ankle brachial index (ABI) <=0.90 at the baseline study visit is an inclusion criterion for PAD.
* Second, potential participants who have an ABI > 0.90 but ≤ 1.00 and experience a 20% or higher drop in ABI after heel-rise exercise will be eligible.
* Third, potential participants with an ABI > 0.90 who have vascular lab evidence of PAD or angiographic evidence of PAD who have ischemic symptoms during the six-minute walk and/or treadmill exercise stress test will be eligible.
* Fourth, potential participants with a history of lower extremity revascularization who do not meet the criterion above and have an ABI > 0.90 with a 20% or higher drop in ABI after heel-rise exercise will be eligible.

Exclusion Criteria:

* Above- or below-knee amputation.
* Critical limb ischemia.
* Wheelchair-bound or requiring a walker to ambulate.
* Walking is limited by a symptom other than PAD.
* Current foot ulcer on bottom of foot.
* Diabetes mellitus defined as one or more of a) patient report of physician diagnosed diabetes mellitus, b) use of one or more diabetes medications, c) two baseline hemoglobinA1C values of >6.5, d) two fasting glucose values >126 mg/dl. [NOTE: the second fasting glucose value and hemoglobin A1C values will be at the discretion of the principal investigator. For example, if the first glucose value is >300 or the first A1C value is >6.9, then investigators may decide not to repeat the value.]
* Chronic kidney disease defined as GFR <=45. [NOTE: if GFR is 40-44, investigator discretion will be used to determine if a repeat test may be performed. If the second GFR value is >45, the participant may be included.]
* Chronic liver disease defined as two or more hepatic function tests >=2.0 times the upper limit of normal. [NOTE: participants who meet this criterion may undergo a re-test of hepatic function tests to determine whether initially elevated hepatic enzymes represented a transient or spurious phenomenon.]
* Failure to successfully complete the 2-week study run-in, defined as unable to tolerate metformin and/or failing to take the medication daily for 10 or more days in the two-week period.
* Planned lower extremity revascularization, orthopedic surgery, or other major surgery during the next six months.
* Lower extremity revascularization, orthopedic surgery, cardiovascular event, coronary revascularization, or other major surgery in the previous three months.
* Major medical illness including renal disease requiring dialysis, lung disease requiring oxygen, Parkinson's disease, a life-threatening illness with life expectancy less than six months, or cancer requiring treatment in the previous two years. [NOTE: potential participants may still qualify if they have had treatment for an early stage cancer in the past two years and the prognosis is excellent. Participants who only use oxygen at night may still qualify.]
* Mini-Mental Status Examination (MMSE) score <23 or dementia. However, investigator discretion may be used to allow some people below this threshold to participate, if the investigator determines there is another reason for their lower score, including lack of familiarity with the English language or lack of sufficient education to achieve a score of 23 or higher. Note that the MMSE include some spelling and English writing proficiency.
* Participation in or completion of a clinical trial in the previous three months. [NOTE: after completing a stem cell or gene therapy intervention, participants will become eligible after the final study follow-up visit of the stem cell or gene therapy study so long as at least six months have passed since the final intervention administration. After completing a supplement or drug therapy (other than stem cell or gene therapy), participants will be eligible after the final study follow-up visit as long as at least three months have passed since the final intervention of the trial.]
* Currently taking metformin or has taken metformin in past six months.
* Increase in angina or angina at rest
* Non-English speaking.
* Visual impairment that limits walking ability.
* In addition to the above criteria, investigator discretion will be used to determine if the trial is unsafe or not a good fit for the potential participant.

Vulnerable populations (fetuses, pregnant women, children, prisoners, and institutionalized persons) and adults unable to consent will not be included in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 203 (Actual)
Dates: Start 2017-05-23 (Actual); Primary Completion 2025-08-20 (Actual); Study Completion 2025-11 (Estimated)

PRIMARY OUTCOMES:
Six-minute walk performance | Change from baseline to six-month follow-up
  Participants walking up and down a 100 foot hallway for six minutes following a standardized protocol. The goal is for them to walk as far as possible in six minutes

SECONDARY OUTCOMES:
Maximal treadmill walking time | Change from baseline to six-month follow-up
  A Gardner treadmill exercise protocol will be used
Brachial artery flow-mediated dilation | Change from baseline to six-month follow-up
  Upper brachial artery flow-mediated dilation will be assessed using a standard protocol
The Walking Impairment Questionnaire | Change from baseline to six-month follow-up
  The well validated Walking Impairment Questionnaire will be used to measure patient- perceived walking performance.
The SF-36 Physical Functioning Score | Change from baseline to six-month follow-up
  This well validated quality of life measure will be used to assess changes in patient perceived quality of life.
Calf muscle biopsy biochemical measures | Change from baseline to six-month follow-up
  A skeletal muscle sample will be obtained from the gastrocnemius muscle.

CONTACTS AND LOCATIONS:
Overall Officials: Mary McDermott, MD, Principal Investigator — Northwestern University
Locations (5):
- United States (5):
  - University of Florida, Gainesville, Florida
  - Northwestern University, Chicago, Illinois
  - University of Chicago, Chicago, Illinois
  - Tulane University, New Orleans, Louisiana
  - Ochsner Medical Center, New Orleans, Louisiana

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] McDermott MM, Domanchuk KJ, Tian L, Zhao L, Zhang D, Bazzano L, Berceli S, Criqui MH, Ferrucci L, Guralnik JM, Leeuwenburgh C, Ho KJ, Ismaeel A, Kibbe MR, Korcarz C, Kosmac K, Lloyd-Jones D, Peterson CA, Stein JH, Sufit R, Wilkins J, Polonsky TS. Metformin to Improve Walking Performance in Lower Extremity Peripheral Artery Disease: The PERMET Randomized Clinical Trial. JAMA. 2026 Feb 3;335(5):407-415. doi: 10.1001/jama.2025.21358. PMID 41205146
- [Derived] Nayak P, Polonsky T, Tian L, Greenland P, Xu S, Zhang D, Zhao L, Criqui MH, Kibbe MR, Gladders B, Goodney P, Ho K, Guralnik JM, McDermott MM. Medical therapies, comorbid conditions, and functional performance in people with peripheral artery disease enrolled in clinical trials between 2004 and 2021. Vasc Med. 2023 Apr;28(2):144-146. doi: 10.1177/1358863X221145533. Epub 2023 Jan 1. PMID 36588397